CLINICAL TRIAL: NCT03328845
Title: Impact on the Oxidative Stress of the Different Analogues of Insulin in People With Type 1 Diabetes. Clinical Trial of Low Level of Intervention. (Ineox Study)
Brief Title: Impact on the Oxidative Stress of the Different Analogues of Insulin in People With Type 1 Diabetes. (Ineox Study)
Acronym: INEOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Principal Investigator, Virginia Morillas, Maria Soledad Ruiz de Adana, Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIM-EOX-2016-01
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Oxidation; Insulin analogues; Type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Lispro; Insulin Aspart; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Tresiba & NovoRapid (Other): Patients treated with Tresiba insulin and NovoRapid insulin
  Interventions: Drug: Tresiba; Drug: NovoRapid
- Toujeo SoloStar & NovoRapid (Other): Patients treated with Toujeo SoloStar insulin and NovoRapid insulin
  Interventions: Drug: Toujeo SoloStar; Drug: NovoRapid
- Tresiba & Humalog Kwikpen (Other): Patients treated with Tresiba insulin and Humalog kwikpen insulin
  Interventions: Drug: Tresiba; Drug: Humalog Kwikpen
- Toujeo SoloStar & Humalog Kwikpen (Other): Patients treated with Toujeo SoloStar insulin and Humalog kwikpen insulin
  Interventions: Drug: Toujeo SoloStar; Drug: Humalog Kwikpen
- Tresiba & Apidra (Other): Patients treated with Tresiba insulin and Apidra insulin
  Interventions: Drug: Tresiba; Drug: Apidra
- Toujeo SoloStar & Apidra (Other): Patients treated with Toujeo SoloStar insulin and Apidra insulin
  Interventions: Drug: Toujeo SoloStar; Drug: Apidra

INTERVENTIONS:
Drug: Toujeo SoloStar — Basal insulin at 16.00h and optimization of this basal doses with objetives of glycaemia before breakfast betwen 80-130 mg/ dl.
  Other Names: Glargina U300
  Arms: Toujeo SoloStar & Apidra; Toujeo SoloStar & Humalog Kwikpen; Toujeo SoloStar & NovoRapid
Drug: Tresiba — Basal insulin at 16.00h and optimization of this basal doses with objetives of glycaemia before breakfast betwen 80-130 mg/ dl.
  Other Names: Degludec insulin
  Arms: Tresiba & Apidra; Tresiba & Humalog Kwikpen; Tresiba & NovoRapid
Drug: Humalog Kwikpen — Ultrarrapid insulin that the patient had already and dose adjustement to obtain postprandial glycaemia levels < 150 mg/dl
  Other Names: Lispro insulin
  Arms: Toujeo SoloStar & Humalog Kwikpen; Tresiba & Humalog Kwikpen
Drug: NovoRapid — Ultrarrapid insulin that the patient had already and dose adjustement to obtain postprandial glycaemia levels < 150 mg/dl
  Other Names: Aspart insulin
  Arms: Toujeo SoloStar & NovoRapid; Tresiba & NovoRapid
Drug: Apidra — Ultrarrapid insulin that the patient had already and dose adjustement to obtain postprandial glycaemia levels < 150 mg/dl
  Other Names: Glulisine insulin
  Arms: Toujeo SoloStar & Apidra; Tresiba & Apidra

SUMMARY:
This study evaluates in a group of people with DM 1 the influence in parameters of oxidative stress of the treatments with the different current analogs of insulin

DETAILED DESCRIPTION:
To evaluate by a randomized study in a group of people with DM 1 the influence in parameters of oxidative stress of the treatments with the different current analogs of

Insulin by analyzing:

1. - The circulating levels of oxidative stress markers: A) Anti oxidation: Total antioxidant capacity (CAT), B) Oxidation: 8-iso-prostaglandin F2 alpha (8-iso-PGF2α), acid reactive substances Thiobarbituric (TBARS) and LDL-oxidized.
2. - The relationship between glycemic control variables (HbA1c and mean glycemia) and variability (Standard deviation (SD), coefficient of variation (CV), and MAGE (mean amplitude of Glycemic excursions) and oxidative stress parameters analyzed.

Goal 2:

Study the activation of cellular pathways associated with processes and oxidation states, by means of a Array of expression of up to 50 genes encoding oxidative stress response genes as CPT1a (Carnitine Palmitoyl Transferase 1a, mitochondrial oxidizing b limiting enzyme), TAS (Fatty acyl synthetase), acetyl-coA carboxylase, Acadm (medium chain acyl dehydrogenase), Acadl (long chain acyl dehydrogenase), Acadvl (long chain acyl coA dehydrogenase), SOD1, Hmox1 and Glutamine-Cysteine ligase (Gclc).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 65 years (inclusive).
* DM1 of more than two years of evolution with habitual follow-up in the Diabetes Unit of the University Regional Hospital of Malaga.
* HbA1c ≤ 10%
* Intensive treatment with basal MDI - Bowl for more than 12 months prior to the start of study.
* Gives informed consent.

Exclusion Criteria:

* Chronic kidney disease, liver disease, thyroid dysfunction (except hypothyroidism correctly treated and controlled).
* Pregnancy or pregnancy planning.
* Diabetes mellitus type 2.
* Hyperuricemia (uric acid ≥7 mg / dl at the time of inclusion or current treatment With allopurinol).
* Absence of collaboration (informed consent).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Oxidative stress markers with the new slow insulin analogues | 6 month
  To evaluate the impact on the circulating levels of oxidative stress markers of the different treatments using the new slow insulin analogues. 1a) Anti oxidation: Total antioxidant capacity (CAT), and 1b) Oxidation: 8-iso-prostaglandin F2 alpha (8-iso-PGF2α), thiobarbituric acid reactive substances (TBARS) and LDL-oxidized

SECONDARY OUTCOMES:
HbA1c | 6 month
  Glycemic control: glycosylated hemoglobin
Mean blood glucose | 6 month
  Glycemic control: mean blood glucose (mg/dl)
Standard deviation | 6 month
  Glycemic variability :standard deviation [SD]
Number of mild hypoglycemia | 6 month
  Number of mild hypoglycaemia in two weeks
Number of severe hypoglycemia | 6 month
  Number of severe hypoglycemia in the last 6 months
Number of hyperglycemia | 6 month
  Number of hyperglycemia> 250 mg / dl in two weeks
Episodes of ketosis | 6 month
  Episodes of ketosis in the last 6 months
Number os hospital admissions | 6 month
  Number of hospital admissions for acute diabetes decompensation in the last 6 months.
Quality of life questionnaire in diabetes (DQOL) | 6 month
  34 items on the quality of life of people with type 1 diabetes
Scale of adherence to treatment in patients with diabetes type 1 (DM1) | 6 month
  15 items related to adherence to patient treatment
Diabetes distress scale. DDS | 6 month
  17 items on the problems and stress that people with type 1 diabetes suffer (Polonski y col, 2005)
Fear of hypoglycemia: Questionnaire FH-15 | 6 month
  15 items related to the fear of hypoglycemia in patients with type 1 diabetes
Diabetes treatment satisfaction questionnaire (DTSQ). | 6 month
  8 items concerning the satisfaction of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Regional University Hospital of Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aljada A, Ghanim H, Saadeh R, Dandona P. Insulin inhibits NFkappaB and MCP-1 expression in human aortic endothelial cells. J Clin Endocrinol Metab. 2001 Jan;86(1):450-3. doi: 10.1210/jcem.86.1.7278. PMID 11232040
- [Background] Arufe MC, Lu M, Lin RY. Differentiation of murine embryonic stem cells to thyrocytes requires insulin and insulin-like growth factor-1. Biochem Biophys Res Commun. 2009 Apr 3;381(2):264-70. doi: 10.1016/j.bbrc.2009.02.035. Epub 2009 Feb 14. PMID 19232325
- [Background] Bashan N, Kovsan J, Kachko I, Ovadia H, Rudich A. Positive and negative regulation of insulin signaling by reactive oxygen and nitrogen species. Physiol Rev. 2009 Jan;89(1):27-71. doi: 10.1152/physrev.00014.2008. PMID 19126754
- [Background] Baynes JW. Role of oxidative stress in development of complications in diabetes. Diabetes. 1991 Apr;40(4):405-12. doi: 10.2337/diab.40.4.405. PMID 2010041
- [Background] Baynes JW, Thorpe SR. Role of oxidative stress in diabetic complications: a new perspective on an old paradigm. Diabetes. 1999 Jan;48(1):1-9. doi: 10.2337/diabetes.48.1.1. PMID 9892215
- [Background] Berg TJ, Nourooz-Zadeh J, Wolff SP, Tritschler HJ, Bangstad HJ, Hanssen KF. Hydroperoxides in plasma are reduced by intensified insulin treatment. A randomized controlled study of IDDM patients with microalbuminuria. Diabetes Care. 1998 Aug;21(8):1295-300. doi: 10.2337/diacare.21.8.1295. PMID 9702436
- [Background] Bergenstal RM, Bailey TS, Rodbard D, Ziemen M, Guo H, Muehlen-Bartmer I, Ahmann AJ. Comparison of Insulin Glargine 300 Units/mL and 100 Units/mL in Adults With Type 1 Diabetes: Continuous Glucose Monitoring Profiles and Variability Using Morning or Evening Injections. Diabetes Care. 2017 Apr;40(4):554-560. doi: 10.2337/dc16-0684. Epub 2017 Jan 23. PMID 28115474
- [Background] Bode BW, Buse JB, Fisher M, Garg SK, Marre M, Merker L, Renard E, Russell-Jones DL, Hansen CT, Rana A, Heller SR; BEGIN(R) Basal-Bolus Type 1 trial investigators. Insulin degludec improves glycaemic control with lower nocturnal hypoglycaemia risk than insulin glargine in basal-bolus treatment with mealtime insulin aspart in Type 1 diabetes (BEGIN((R)) Basal-Bolus Type 1): 2-year results of a randomized clinical trial. Diabet Med. 2013 Nov;30(11):1293-7. doi: 10.1111/dme.12243. Epub 2013 Jun 17. PMID 23710902
- [Background] Bravi MC, Armiento A, Laurenti O, Cassone-Faldetta M, De Luca O, Moretti A, De Mattia G. Insulin decreases intracellular oxidative stress in patients with type 2 diabetes mellitus. Metabolism. 2006 May;55(5):691-5. doi: 10.1016/j.metabol.2006.01.003. PMID 16631447
- [Background] Brownlee M. The pathobiology of diabetic complications: a unifying mechanism. Diabetes. 2005 Jun;54(6):1615-25. doi: 10.2337/diabetes.54.6.1615. No abstract available. PMID 15919781
- [Background] Ceolotto G, Bevilacqua M, Papparella I, Baritono E, Franco L, Corvaja C, Mazzoni M, Semplicini A, Avogaro A. Insulin generates free radicals by an NAD(P)H, phosphatidylinositol 3'-kinase-dependent mechanism in human skin fibroblasts ex vivo. Diabetes. 2004 May;53(5):1344-51. doi: 10.2337/diabetes.53.5.1344. PMID 15111505
- [Background] Ceriello A. Hyperglycaemia and the vessel wall: the pathophysiological aspects on the atherosclerotic burden in patients with diabetes. Eur J Cardiovasc Prev Rehabil. 2010 May;17 Suppl 1:S15-9. doi: 10.1097/01.hjr.0000368193.24732.66. PMID 20489415
- [Background] Ceriello A, Esposito K, Ihnat M, Thorpe J, Giugliano D. Effect of acute hyperglycaemia, long-term glycaemic control and insulin on endothelial dysfunction and inflammation in Type 1 diabetic patients with different characteristics. Diabet Med. 2010 Aug;27(8):911-7. doi: 10.1111/j.1464-5491.2009.02928.x. PMID 20653749
- [Background] Ceriello A, Ihnat M. Oxidative stress is, convincingly, the mediator of the dangerous effects of glucose variability. Diabet Med. 2010 Aug;27(8):968. doi: 10.1111/j.1464-5491.2010.02931.x. No abstract available. PMID 20653758
- [Background] Ceriello A, Novials A, Ortega E, Canivell S, La Sala L, Pujadas G, Esposito K, Giugliano D, Genovese S. Glucagon-like peptide 1 reduces endothelial dysfunction, inflammation, and oxidative stress induced by both hyperglycemia and hypoglycemia in type 1 diabetes. Diabetes Care. 2013 Aug;36(8):2346-50. doi: 10.2337/dc12-2469. Epub 2013 Apr 5. PMID 23564922
- [Background] Costacou T, Evans RW, Schafer GL, Orchard TJ. Oxidative stress and response in relation to coronary artery disease in type 1 diabetes. Diabetes Care. 2013 Nov;36(11):3503-9. doi: 10.2337/dc12-2378. Epub 2013 Aug 6. PMID 23920084
- [Background] Costacou T, Lopes-Virella MF, Zgibor JC, Virella G, Otvos J, Walsh M, Orchard TJ. Markers of endothelial dysfunction in the prediction of coronary artery disease in type 1 diabetes. The Pittsburgh Epidemiology of Diabetes Complications Study. J Diabetes Complications. 2005 Jul-Aug;19(4):183-93. doi: 10.1016/j.jdiacomp.2005.01.003. PMID 15993351
- [Background] Chang L, Chiang SH, Saltiel AR. Insulin signaling and the regulation of glucose transport. Mol Med. 2004 Jul-Dec;10(7-12):65-71. doi: 10.2119/2005-00029.Saltiel. PMID 16307172
- [Background] Dandona P, Aljada A, Mohanty P, Ghanim H, Hamouda W, Assian E, Ahmad S. Insulin inhibits intranuclear nuclear factor kappaB and stimulates IkappaB in mononuclear cells in obese subjects: evidence for an anti-inflammatory effect? J Clin Endocrinol Metab. 2001 Jul;86(7):3257-65. doi: 10.1210/jcem.86.7.7623. PMID 11443198
- [Background] Dandona P, Chaudhuri A, Ghanim H, Mohanty P. Effect of hyperglycemia and insulin in acute coronary syndromes. Am J Cardiol. 2007 Jun 4;99(11A):12H-18H. doi: 10.1016/j.amjcard.2007.04.004. PMID 17665748
- [Background] Dandona P, Chaudhuri A, Ghanim H, Mohanty P. Insulin as an anti-inflammatory and antiatherogenic modulator. J Am Coll Cardiol. 2009 Feb 3;53(5 Suppl):S14-20. doi: 10.1016/j.jacc.2008.10.038. PMID 19179212
- [Background] Davies MJ, Derezinski T, Pedersen CB, Clauson P. Reduced weight gain with insulin detemir compared to NPH insulin is not explained by a reduction in hypoglycemia. Diabetes Technol Ther. 2008 Aug;10(4):273-7. doi: 10.1089/dia.2008.0282. PMID 18715200
- [Background] Weight gain associated with intensive therapy in the diabetes control and complications trial. The DCCT Research Group. Diabetes Care. 1988 Jul-Aug;11(7):567-73. doi: 10.2337/diacare.11.7.567. PMID 2904881
- [Background] Dominguez C, Ruiz E, Gussinye M, Carrascosa A. Oxidative stress at onset and in early stages of type 1 diabetes in children and adolescents. Diabetes Care. 1998 Oct;21(10):1736-42. doi: 10.2337/diacare.21.10.1736. PMID 9773740
- [Background] Fawcett J, Tsui BT, Kruer MC, Duckworth WC. Reduced action of insulin glargine on protein and lipid metabolism: possible relationship to cellular hormone metabolism. Metabolism. 2004 Aug;53(8):1037-44. doi: 10.1016/j.metabol.2004.02.013. PMID 15281015
- [Background] Francescato MP, Stel G, Geat M, Cauci S. Oxidative stress in patients with type 1 diabetes mellitus: is it affected by a single bout of prolonged exercise? PLoS One. 2014 Jun 6;9(6):e99062. doi: 10.1371/journal.pone.0099062. eCollection 2014. PMID 24905823
- [Background] Franklin VL, Khan F, Kennedy G, Belch JJ, Greene SA. Intensive insulin therapy improves endothelial function and microvascular reactivity in young people with type 1 diabetes. Diabetologia. 2008 Feb;51(2):353-60. doi: 10.1007/s00125-007-0870-2. Epub 2007 Nov 27. PMID 18040663
- [Background] Garcia-Escobar E, Rodriguez-Pacheco F, Haro-Mora JJ, Gomez-Zumaquero JM, Rubio-Martin E, Gutierrez-Repiso C, Soriguer F, Rojo-Martinez G. Effect of insulin analogues on 3t3-l1 adipogenesis and lipolysis. Eur J Clin Invest. 2011 Sep;41(9):979-86. doi: 10.1111/j.1365-2362.2011.02492.x. Epub 2011 Mar 2. PMID 21366560
- [Background] Giacco F, Brownlee M. Oxidative stress and diabetic complications. Circ Res. 2010 Oct 29;107(9):1058-70. doi: 10.1161/CIRCRESAHA.110.223545. PMID 21030723
- [Background] Goldman J, White JR Jr. New Insulin Glargine 300 U/mL for the Treatment of Type 1 and Type 2 Diabetes Mellitus. Ann Pharmacother. 2015 Oct;49(10):1153-61. doi: 10.1177/1060028015597915. Epub 2015 Aug 3. PMID 26238470
- [Background] Heinemann L, Linkeschova R, Rave K, Hompesch B, Sedlak M, Heise T. Time-action profile of the long-acting insulin analog insulin glargine (HOE901) in comparison with those of NPH insulin and placebo. Diabetes Care. 2000 May;23(5):644-9. doi: 10.2337/diacare.23.5.644. PMID 10834424
- [Background] Heise T, Hermanski L, Nosek L, Feldman A, Rasmussen S, Haahr H. Insulin degludec: four times lower pharmacodynamic variability than insulin glargine under steady-state conditions in type 1 diabetes. Diabetes Obes Metab. 2012 Sep;14(9):859-64. doi: 10.1111/j.1463-1326.2012.01627.x. Epub 2012 Jun 7. PMID 22594461
- [Background] Home PD, Bergenstal RM, Bolli GB, Ziemen M, Rojeski M, Espinasse M, Riddle MC. New Insulin Glargine 300 Units/mL Versus Glargine 100 Units/mL in People With Type 1 Diabetes: A Randomized, Phase 3a, Open-Label Clinical Trial (EDITION 4). Diabetes Care. 2015 Dec;38(12):2217-25. doi: 10.2337/dc15-0249. Epub 2015 Jun 17. PMID 26084341
- [Background] Hoeldtke RD, Bryner KD, Hoeldtke ME, Christie I, Ganser G, Hobbs G, Riggs J. Sympathetic sudomotor disturbance in early type 1 diabetes mellitus is linked to lipid peroxidation. Metabolism. 2006 Nov;55(11):1524-31. doi: 10.1016/j.metabol.2006.06.023. PMID 17046556
- [Background] Homko C, Deluzio A, Jimenez C, Kolaczynski JW, Boden G. Comparison of insulin aspart and lispro: pharmacokinetic and metabolic effects. Diabetes Care. 2003 Jul;26(7):2027-31. doi: 10.2337/diacare.26.7.2027. PMID 12832307
- [Background] Liu HY, Cao SY, Hong T, Han J, Liu Z, Cao W. Insulin is a stronger inducer of insulin resistance than hyperglycemia in mice with type 1 diabetes mellitus (T1DM). J Biol Chem. 2009 Oct 2;284(40):27090-100. doi: 10.1074/jbc.M109.016675. Epub 2009 Aug 4. PMID 19654321
- [Background] Hojlund K, Poulsen M, Staehr P, Brusgaard K, Beck-Nielsen H. Effect of insulin on protein phosphatase 2A expression in muscle in type 2 diabetes. Eur J Clin Invest. 2002 Dec;32(12):918-23. doi: 10.1046/j.1365-2362.2002.01098.x. PMID 12534451
- [Background] Jarvisalo MJ, Raitakari M, Toikka JO, Putto-Laurila A, Rontu R, Laine S, Lehtimaki T, Ronnemaa T, Viikari J, Raitakari OT. Endothelial dysfunction and increased arterial intima-media thickness in children with type 1 diabetes. Circulation. 2004 Apr 13;109(14):1750-5. doi: 10.1161/01.CIR.0000124725.46165.2C. Epub 2004 Mar 15. PMID 15023875
- [Background] Kalra S, Baruah MP, Niazi AK. Degludec: a novel basal insulin. Recent Pat Endocr Metab Immune Drug Discov. 2012 Jan;6(1):18-23. doi: 10.2174/187221412799015326. PMID 22280221
- [Background] Korytkowski MT, Salata RJ, Koerbel GL, Selzer F, Karslioglu E, Idriss AM, Lee KK, Moser AJ, Toledo FG. Insulin therapy and glycemic control in hospitalized patients with diabetes during enteral nutrition therapy: a randomized controlled clinical trial. Diabetes Care. 2009 Apr;32(4):594-6. doi: 10.2337/dc08-1436. PMID 19336639
- [Background] Kurtzhals P, Schaffer L, Sorensen A, Kristensen C, Jonassen I, Schmid C, Trub T. Correlations of receptor binding and metabolic and mitogenic potencies of insulin analogs designed for clinical use. Diabetes. 2000 Jun;49(6):999-1005. doi: 10.2337/diabetes.49.6.999. PMID 10866053
- [Background] Laaksonen DE, Atalay M, Niskanen L, Uusitupa M, Hanninen O, Sen CK. Increased resting and exercise-induced oxidative stress in young IDDM men. Diabetes Care. 1996 Jun;19(6):569-74. doi: 10.2337/diacare.19.6.569. PMID 8725853
- [Background] Lepore M, Pampanelli S, Fanelli C, Porcellati F, Bartocci L, Di Vincenzo A, Cordoni C, Costa E, Brunetti P, Bolli GB. Pharmacokinetics and pharmacodynamics of subcutaneous injection of long-acting human insulin analog glargine, NPH insulin, and ultralente human insulin and continuous subcutaneous infusion of insulin lispro. Diabetes. 2000 Dec;49(12):2142-8. doi: 10.2337/diabetes.49.12.2142. PMID 11118018
- [Background] Liebl A, Prager R, Binz K, Kaiser M, Bergenstal R, Gallwitz B; PREFER Study Group. Comparison of insulin analogue regimens in people with type 2 diabetes mellitus in the PREFER Study: a randomized controlled trial. Diabetes Obes Metab. 2009 Jan;11(1):45-52. doi: 10.1111/j.1463-1326.2008.00915.x. Epub 2008 Jul 17. PMID 18643839
- [Background] Makimattila S, Virkamaki A, Malmstrom R, Utriainen T, Yki-Jarvinen H. Insulin resistance in type I diabetes mellitus: a major role for reduced glucose extraction. J Clin Endocrinol Metab. 1996 Feb;81(2):707-12. doi: 10.1210/jcem.81.2.8636292.
- [Background] Mannucci E, Monami M, Marchionni N. Short-acting insulin analogues vs. regular human insulin in type 2 diabetes: a meta-analysis. Diabetes Obes Metab. 2009 Jan;11(1):53-9. doi: 10.1111/j.1463-1326.2008.00934.x. Epub 2008 Jul 29. PMID 18671795
- [Background] Marra G, Cotroneo P, Pitocco D, Manto A, Di Leo MA, Ruotolo V, Caputo S, Giardina B, Ghirlanda G, Santini SA. Early increase of oxidative stress and reduced antioxidant defenses in patients with uncomplicated type 1 diabetes: a case for gender difference. Diabetes Care. 2002 Feb;25(2):370-5. doi: 10.2337/diacare.25.2.370. PMID 11815512
- [Background] Matsuhisa M, Koyama M, Cheng X, Sumi M, Riddle MC, Bolli GB, Hirose T; EDITION JP 1 study group. Sustained glycaemic control and less nocturnal hypoglycaemia with insulin glargine 300U/mL compared with glargine 100U/mL in Japanese adults with type 1 diabetes (EDITION JP 1 randomised 12-month trial including 6-month extension). Diabetes Res Clin Pract. 2016 Dec;122:133-140. doi: 10.1016/j.diabres.2016.10.002. Epub 2016 Oct 13. PMID 27835765
- [Background] Delmastro MM, Piganelli JD. Oxidative stress and redox modulation potential in type 1 diabetes. Clin Dev Immunol. 2011;2011:593863. doi: 10.1155/2011/593863. Epub 2011 May 18. PMID 21647409
- [Background] Monnier L, Colette C, Mas E, Michel F, Cristol JP, Boegner C, Owens DR. Regulation of oxidative stress by glycaemic control: evidence for an independent inhibitory effect of insulin therapy. Diabetologia. 2010 Mar;53(3):562-71. doi: 10.1007/s00125-009-1574-6. Epub 2009 Nov 5. PMID 19890623
- [Background] Monnier L, Hanefeld M, Schnell O, Colette C, Owens D. Insulin and atherosclerosis: how are they related? Diabetes Metab. 2013 Apr;39(2):111-7. doi: 10.1016/j.diabet.2013.02.001. Epub 2013 Mar 15. PMID 23507269
- [Background] Muchmore DB, Heinemann L, Tamborlane W, Wu XW, Fleming A. Assessing rates of hypoglycemia as an end point in clinical trials. Diabetes Care. 2015 Oct;38(10):e160-1. doi: 10.2337/dc15-0808. Epub 2015 Aug 17. No abstract available. PMID 26283738
- [Background] Muretta JM, Mastick CC. How insulin regulates glucose transport in adipocytes. Vitam Horm. 2009;80:245-86. doi: 10.1016/S0083-6729(08)00610-9. PMID 19251041
- [Background] Nandish S, Wyatt J, Bailon O, Smith M, Oliveros R, Chilton R. Implementing cardiovascular risk reduction in patients with cardiovascular disease and diabetes mellitus. Am J Cardiol. 2011 Aug 2;108(3 Suppl):42B-51B. doi: 10.1016/j.amjcard.2011.03.015. PMID 21802580
- [Background] ORIGIN Trial Investigators; Gerstein HC, Bosch J, Dagenais GR, Diaz R, Jung H, Maggioni AP, Pogue J, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. Basal insulin and cardiovascular and other outcomes in dysglycemia. N Engl J Med. 2012 Jul 26;367(4):319-28. doi: 10.1056/NEJMoa1203858. Epub 2012 Jun 11. PMID 22686416
- [Background] Osterberg O, Erichsen L, Ingwersen SH, Plum A, Poulsen HE, Vicini P. Pharmacokinetic and pharmacodynamic properties of insulin aspart and human insulin. J Pharmacokinet Pharmacodyn. 2003 Jun;30(3):221-35. doi: 10.1023/a:1025594110558. PMID 14571692
- [Background] Scheen AJ. New therapeutic approaches in type 2 diabetes. Acta Clin Belg. 2008 Nov-Dec;63(6):402-7. doi: 10.1179/acb.2008.083. PMID 19170358
- [Background] Razavi Nematollahi L, Kitabchi AE, Stentz FB, Wan JY, Larijani BA, Tehrani MM, Gozashti MH, Omidfar K, Taheri E. Proinflammatory cytokines in response to insulin-induced hypoglycemic stress in healthy subjects. Metabolism. 2009 Apr;58(4):443-8. doi: 10.1016/j.metabol.2008.10.018. PMID 19303962
- [Background] Rosenstock J, Dailey G, Massi-Benedetti M, Fritsche A, Lin Z, Salzman A. Reduced hypoglycemia risk with insulin glargine: a meta-analysis comparing insulin glargine with human NPH insulin in type 2 diabetes. Diabetes Care. 2005 Apr;28(4):950-5. doi: 10.2337/diacare.28.4.950. PMID 15793205
- [Background] Sanders EJ, Harvey S. Peptide hormones as developmental growth and differentiation factors. Dev Dyn. 2008 Jun;237(6):1537-52. doi: 10.1002/dvdy.21573. PMID 18498096
- [Background] Seaquist ER, Anderson J, Childs B, Cryer P, Dagogo-Jack S, Fish L, Heller SR, Rodriguez H, Rosenzweig J, Vigersky R. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013 May;36(5):1384-95. doi: 10.2337/dc12-2480. Epub 2013 Apr 15. PMID 23589542
- [Background] Singh P, Jain A, Kaur G. Impact of hypoglycemia and diabetes on CNS: correlation of mitochondrial oxidative stress with DNA damage. Mol Cell Biochem. 2004 May;260(1-2):153-9. doi: 10.1023/b:mcbi.0000026067.08356.13. PMID 15228097
- [Background] Somwar R, Sweeney G, Ramlal T, Klip A. Stimulation of glucose and amino acid transport and activation of the insulin signaling pathways by insulin lispro in L6 skeletal muscle cells. Clin Ther. 1998 Jan-Feb;20(1):125-40. doi: 10.1016/s0149-2918(98)80040-4. PMID 9522110
- [Background] Steensgaard DB, Schluckebier G, Strauss HM, Norrman M, Thomsen JK, Friderichsen AV, Havelund S, Jonassen I. Ligand-controlled assembly of hexamers, dihexamers, and linear multihexamer structures by the engineered acylated insulin degludec. Biochemistry. 2013 Jan 15;52(2):295-309. doi: 10.1021/bi3008609. Epub 2013 Jan 3. PMID 23256685
- [Background] Varvarovska J, Racek J, Stetina R, Sykora J, Pomahacova R, Rusavy Z, Lacigova S, Trefil L, Siala K, Stozicky F. Aspects of oxidative stress in children with type 1 diabetes mellitus. Biomed Pharmacother. 2004 Dec;58(10):539-45. doi: 10.1016/j.biopha.2004.09.011. PMID 15589060
- [Background] Vora J, Christensen T, Rana A, Bain SC. Insulin degludec versus insulin glargine in type 1 and type 2 diabetes mellitus: a meta-analysis of endpoints in phase 3a trials. Diabetes Ther. 2014 Dec;5(2):435-46. doi: 10.1007/s13300-014-0076-9. Epub 2014 Aug 1. PMID 25081590
- [Background] Wang J, Alexanian A, Ying R, Kizhakekuttu TJ, Dharmashankar K, Vasquez-Vivar J, Gutterman DD, Widlansky ME. Acute exposure to low glucose rapidly induces endothelial dysfunction and mitochondrial oxidative stress: role for AMP kinase. Arterioscler Thromb Vasc Biol. 2012 Mar;32(3):712-20. doi: 10.1161/ATVBAHA.111.227389. Epub 2011 Dec 29. PMID 22207730
- [Background] Wolff SP, Dean RT. Glucose autoxidation and protein modification. The potential role of 'autoxidative glycosylation' in diabetes. Biochem J. 1987 Jul 1;245(1):243-50. doi: 10.1042/bj2450243. PMID 3117042
- [Background] Wright RJ, Frier BM. Vascular disease and diabetes: is hypoglycaemia an aggravating factor? Diabetes Metab Res Rev. 2008 Jul-Aug;24(5):353-63. doi: 10.1002/dmrr.865. PMID 18461635
- [Background] Zib I, Raskin P. Novel insulin analogues and its mitogenic potential. Diabetes Obes Metab. 2006 Nov;8(6):611-20. doi: 10.1111/j.1463-1326.2005.00567.x. PMID 17026485
- [Background] Ziegler D, Buchholz S, Sohr C, Nourooz-Zadeh J, Roden M. Oxidative stress predicts progression of peripheral and cardiac autonomic nerve dysfunction over 6 years in diabetic patients. Acta Diabetol. 2015 Feb;52(1):65-72. doi: 10.1007/s00592-014-0601-3. Epub 2014 Jun 5. PMID 24898524